CLINICAL TRIAL: NCT03929263
Title: The Dyadic Inter-Brain Signaling (DIBS) Project With Parent-Adolescent Training on Neurofeedback and Synchrony
Brief Title: Parent-Adolescent Training on Neurofeedback and Synchrony
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oklahoma State University Center for Health Sciences (Other)
Collaborators: Oklahoma State University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CHS2017011
Record Dates: First submitted 2019-04-22; First posted 2019-04-26 (Actual); Results first posted 2024-09-24 (Actual); Last update posted 2024-09-24 (Actual); Status verified 2024-06

CONDITIONS: Testing Protocol With Healthy Individuals for Feasibility

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Real-time fMRI neurofeedback (Experimental): All participants will receive neurofeedback from the target region (no sham condition).
  Interventions: Behavioral: Real-time fMRI neurofeedback

INTERVENTIONS:
Behavioral: Real-time fMRI neurofeedback — Participants will attempt to regulate own and/or their partner's brain activation in a specified brain region via real-time fMRI neurofeedback.

SUMMARY:
The study will test a real-time functional magnetic resonance imaging (fMRI) hyperscanning neurofeedback protocol for feasibility with ten mothers and their psychiatrically healthy adolescent daughters, with the eventual goal to test this in a sample of depressed adolescents in a future study.

DETAILED DESCRIPTION:
This study will utilize a rigorous multi-method, multi-informant design to examine the effects of dyadic neurofeedback (dnf) on adolescent brain activation with fMRI hyperscanning. Parents and adolescents will also report on emotion regulation, depressive symptoms, and parenting practices. Data collection procedures will take place at the Laureate Institute for Brain Research (LIBR), which is equipped with two identical scanners that have advanced real-time fMRI systems capable of conducting parallel fMRI hyperscanning, including the capacity for neurofeedback. Parents will complete a phone screen to determine initial eligibility. If initial study criteria are met, a 2-hour in-person lab visit will be scheduled where mothers and daughters will complete consent/assent; diagnostic interviews; surveys on emotion regulation, parenting practices, depression, and anxiety; and additional screening. Survey data will be used for preliminary exploratory analyses. Based on data collected from the screening visit, participants will be invited to participate in the full study: a 4-hour visit where mothers and daughters will complete emotion ratings, mock scanner training, and fMRI tasks individually and together using hyperscanning (scan time = 16 min resting-state [2 runs], 7 min structural MRI, 40 min fMRI tasks, 10 min clinical MRI scans).

ELIGIBILITY:
Inclusion Criteria:

* Eligible for fMRI
* Sufficient English fluency to complete tasks
* BMI ≦ 40.0
* Right-handed
* Biological female
* Co-residing at least 4 days/week
* Adult participants: Biological mother of adolescent participant
* Adult participants:Primary caregiver > 50% of child's lifespan
* Adult participants:BMI ≧ 18.0
* Adolescent participants: Age 13-17 years
* Adolescent participants: BMI ≧ 16.0

Exclusion Criteria:

* Current psychiatric diagnosis
* Medications influencing fMRI
* Medical conditions influencing fMRI
* Alcohol or psychoactive drug on scan day
* Adolescent participants: Neurodevelopmental delay
* Adolescent participants: History of mood or psychotic disorder
* Adolescent participants: History of obsessive-compulsive disorder (OCD) or attention-deficit/hyperactivity disorder (ADHD)

Min Age: 13 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2019-09-25 (Actual); Primary Completion 2021-02-27 (Actual); Study Completion 2021-02-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kara L Kerr, PhD, Principal Investigator — Oklahoma State University
Locations (1):
- Laureate Institute for Brain Research, Tulsa, Oklahoma, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kerr KL, Ratliff EL, Cohen ZP, Fuller S, Cosgrove KT, DeVille DC, Misaki M, Morris AS, Bodurka J. Real-Time Functional Magnetic Resonance Imaging Dyadic Neurofeedback for Emotion Regulation: A Proof-of-Concept Study. Front Hum Neurosci. 2022 May 26;16:910951. doi: 10.3389/fnhum.2022.910951. eCollection 2022. PMID 35721350

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Real-time fMRI Neurofeedback
Started | 24
Completed | 24
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Real-time fMRI Neurofeedback
Number analyzed (Participants) | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 12
  Between 18 and 65 years | 12
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 21
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 21
  More than one race | 2
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 24

OUTCOME MEASURES:

1. Primary Outcome: Neurofeedback Rating Scale
Description: Rating scale of perceived effectiveness in completing the task and changing brain activation. Likert scale ranging from 0-10, with higher numbers indicating greater perceived effectiveness.
Time Frame: Baseline (Acquired during scan session)
Population: Parents who participated in at least one neurofeedback session with available data for this outcome variable
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Real-time fMRI Neurofeedback
Number analyzed (Participants) | 11
units on a scale | 5.7 (2.14)

2. Primary Outcome: Emotion Rating Scale
Description: Rating scale asking about current experience of various emotions (happy, sad, angry, etc.). Scale ranges from 0-10, with higher numbers indicating more intense emotions.
Time Frame: Baseline (Acquired during scan session)
Population: Only data from participants used in the neuroimaging results were analyzed.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Real-time fMRI Neurofeedback
Number analyzed (Participants) | 6
units on a scale | 2.11 (1.46)

3. Primary Outcome: Blood Oxygen Level-Dependent (BOLD) Signal Changes (Brain Activation)
Description: Activation in the brain region targeted for neurofeedback and associated regions; resting-state network activity
Time Frame: Baseline (Acquired during scan session)
Population: Only adolescents' data that passed quality control were analyzed. Values are taken from the anterior insula and averaged across scanning runs and participants.
Measure: Mean (Standard Deviation); unit: percent signal change
Arm/Group | Real-time fMRI Neurofeedback
Number analyzed (Participants) | 6
percent signal change | 0.15 (0.38)

ADVERSE EVENTS:
Time Frame: 3 months (Participants completed baseline measures over the course of approximately 1 month followed by 2 months of biweekly follow-ups.)
Description: Definition does not differ from clinicaltrials.gov
Arm/Group | Real-time fMRI Neurofeedback
All-Cause Mortality (participants affected / at risk) | 0/24
Serious Adverse Events (participants affected / at risk) | 0/24
Other Adverse Events (participants affected / at risk) | 0/24

LIMITATIONS AND CAVEATS:
This is a feasibility study with a small sample and no control group.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-03-15): https://cdn.clinicaltrials.gov/large-docs/63/NCT03929263/Prot_SAP_000.pdf
  • Informed Consent Form (2019-05-22): https://cdn.clinicaltrials.gov/large-docs/63/NCT03929263/ICF_001.pdf